CLINICAL TRIAL: NCT03635268
Title: Endophthalmitis After Intravitreal Injection of Antiangiogenic Agents or Corticosteroids, a Cohort Study of the French Population of Patients Who Received Injections Over 9 Years
Acronym: ENIVAC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: MARIET AOI 2017
Record Dates: First submitted 2018-08-14; First posted 2018-08-17 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Intravitreal Injection
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection — Sociodemographic, medical and hospital, on ambulatory care consumption data.

SUMMARY:
Intravitreal injections (IVI) of antiangiogenic agents (AA) have revolutionized the management of age-related macular degeneration (AMD) and diabetic macular edema (DME) in particular. Approximately 600,000 AA IVIs are performed each year in France.

Corticosteroid IVIs are an alternative in the treatment of macular edema when it is diabetic or related to venous occlusion, but also due to inflammation.

Endophthalmitis is one of the most feared complications after IVI because of its poor prognosis, despite its low incidence (values found in the literature between 0.01% and 0.08%). IVI practices have evolved over the years based on the recommendations of specialized organizations, with the current recommendation not to use antibiotic prophylaxis.

The purpose of this study is to study the effect of intravitreal injections of anti-angiogenic agents and corticosteroids on the occurrence of endophthalmitis within 28 days following an injection.

ELIGIBILITY:
Inclusion Criteria:

* adult patients within the French population who had an intravitreal injection, identified by CCAM coding BGLB001
* associated with the delivery of an anti-angiogenic agent or a corticosteroid, identified by the corresponding CIP code
* between February 2007 and November 2015

Exclusion Criteria:

* intraocular surgery less than 42 days before the first injection, identified by the CCAM procedure
* risk factors for endogenous endophthalmitis identified in the 42 days preceding an IVI identified by the ICD10 code

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who has had an intravitreal injection to deliver an anti-angiogenic agent or a corticosteroid
Sampling Method: Non-Probability Sample
Enrollment: 360000 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Frequency of occurrence of endophthalmitis | Up to 28 days following an intravitreal injection

REFERENCES:
- [Result] Baudin F, Benzenine E, Mariet AS, Bron AM, Daien V, Korobelnik JF, Quantin C, Creuzot-Garcher C. Association of Acute Endophthalmitis With Intravitreal Injections of Corticosteroids or Anti-Vascular Growth Factor Agents in a Nationwide Study in France. JAMA Ophthalmol. 2018 Dec 1;136(12):1352-1358. doi: 10.1001/jamaophthalmol.2018.3939. PMID 30242325